CLINICAL TRIAL: NCT01593891
Title: Radiographic and Intravascular (IVUS) Evaluation of Venous Morphology During CCSVI Treatment
Acronym: Resrch_Reg_2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Synergy Health Concepts, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RESEARCH_REGISTRY_2
Record Dates: First submitted 2012-05-06; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: To Determine the Safety and Validity of Venous Angioplasty and; Valvuloplasty in the Treatment of CCSVI. In Addition, it Will; Allow Researchers to Sub-classify Valve Morphology in Relation; to Treatment Success. This Will be Evidenced by Venous Patency; Forty-eight Hours by Doppler Ultrasound as Well as Clinical; Symptom Improvement.
Keywords: IVUS, CCSVI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Radio graphic and Intravascular (IVUS) Evaluation of Venous Morphology During Chronic Cerebral Spinal Venous Insufficiency Treatment

DETAILED DESCRIPTION:
To determine the safety and validity of venous angioplasty and valvuloplasty in the treatment of CCSVI. In addition, it will allow researchers to sub-classify valve morphology in relation to treatment success. This will be evidenced by venous patency forty-eight hours by Doppler ultrasound as well as clinical symptom improvement.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend the nature of the study, including the risks and benefits and execute an informed consent
* Males or Females between the ages of 20 and 60 years of age.
* Voluntary agreement to participate in the study: Radiographic and Intravascular (IVUS) Evaluation of Venous Morphology During CCSVI Treatment.

Exclusion Criteria:

* Any implantable/metallic objects that prevents subject from having a magnetic resonance imaging (MRI/MRV) study.
* History of uncontrolled hypertension
* Previous CCSVI treatment
* Presence of hypercoagulable state
* Special Populations. Special groups include, but are not limited to children, prisoners, pregnant women, fetuses, and cognitively impaired individuals who are unable to provide informed consent.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Many questions remain about how and when CCSVI might play a role in nervous system damage and whether venous angioplasty is helpful in treating the symptoms of CCSVI. Utilizing intravascular ultrasound (IVUS,) this pilot study will provide data that will allow researchers to evaluate venous morphology pre- and post- percutaneous angioplasty and sub-classify valve morphology as related to treatment success by distinguishing vessels which are more responsive to treatment. In addition, this study will validate the safety of valvuloplasty in various neurodegenerative disorders that involve venous obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-08; Study Completion 2012-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Arata, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Synergy Health Concepts Inc., Newport Beach, California, United States